CLINICAL TRIAL: NCT02613364
Title: A Randomized Clinical Trial Comparing the Effectiveness of Yoga, Survivorship Health Education, and Cognitive Behavioral Therapy for Treating Insomnia in Cancer Survivors
Brief Title: Yoga, Survivorship Health Education, and Cognitive Behavioral Therapy in Reducing Insomnia in Cancer Survivors
Acronym: YOCAS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Mustian, Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URCC14040; NCI-2015-01144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RSRB052271 (Other: University of Rochester); URCC14040 (Other: University of Rochester NCORP Research Base); URCC-14040 (Other: DCP); URCC-14040 (Other: CTEP); R01CA181064 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cancer Survivor; Insomnia; Malignant Neoplasm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms | interventions — Behavior Therapy; Early Intervention, Educational; Educational Status; Methods; Monitoring, Physiologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (behavioral intervention-yoga) (Experimental): Patients undergo the YOCAS intervention comprising 18 specific physical postures and mindfulness exercises focused on breathing and meditation and meet with the yoga instructor over 75 minutes 2 times a week for 4 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment
- Arm II (cognitive intervention-CBT-I) (Experimental): Patients undergo CBT-I intervention comprising sleep education, sleep hygiene, sleep restriction, stimulus control, cognitive therapy, and relapse prevention delivered by a health professional over 90 minutes once a week for 8 weeks.
  Interventions: Other: Cognitive Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment
- Arm III (educational intervention) (Active Comparator): Patients attend survivorship health education sessions over 75 minutes 2 times a week for 4 weeks based on the American Society of Clinical Oncology cancer survivorship educational recommendations delivered by a community health educator. Patients also receive a booklet entitled, "Cancer Survivorship Next Steps for Patients and Their Families."
  Interventions: Other: Educational Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment

INTERVENTIONS:
Behavioral: Behavioral Intervention — Undergo yoga intervention
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (behavioral intervention-yoga)
Other: Cognitive Intervention — Undergo CBT-I intervention
  Arms: Arm II (cognitive intervention-CBT-I)
Other: Educational Intervention — Receive health education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm III (educational intervention)
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Monitoring Device — Correlative studies
  Other Names: Monitor
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial compares yoga, survivorship health education program, and cognitive behavioral therapy in reducing sleep disturbance (insomnia) in cancer survivors. Insomnia can be described as excessive daytime napping, difficulty falling asleep, difficulty staying asleep, or waking up earlier than desired. Insomnia can increase fatigue, impair physical function, impair immune function, cause circadian rhythms (known as the biological clock) to be disrupted and decrease quality of life. Yoga may improve circadian rhythms, physical and immune function, and improve insomnia and sleep quality in cancer survivors. It is not yet known whether yoga is more effective at treating insomnia than a health education program or cognitive behavioral therapy program.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if Yoga for Cancer Survivors (YOCAS) is effective for improving patient-reported insomnia (Insomnia Severity Index) compared to Cognitive Behavioral Therapy for Insomnia (CBT-I) and a health education control immediately post intervention.

SECONDARY OBJECTIVES:

I. To examine if YOCAS is effective for improving objective symptoms of insomnia (sleep latency, sleep efficiency, wake after sleep onset, sleep duration, and daytime napping via actigraphy) and global sleep quality impairment (Pittsburgh Sleep Quality Index) compared to CBT-I and a health education control.

II. To examine if YOCAS and CBT-I are effective for maintaining improvements in insomnia (Insomnia Severity Index) 3 and 6 months post intervention compared to a health education control.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients undergo the YOCAS intervention comprising 18 specific physical postures and mindfulness exercises focused on breathing and meditation and meet with the yoga instructor over 75 minutes 2 times a week for 4 weeks.

ARM II: Patients undergo CBT-I intervention comprising sleep education, sleep hygiene, sleep restriction, stimulus control, cognitive therapy, and relapse prevention delivered by a health professional over 90 minutes once a week for 8 weeks.

ARM III: Patients attend survivorship health education sessions over 75 minutes 2 times a week for 4 weeks based on the American Society of Clinical Oncology cancer survivorship educational recommendations delivered by a community health educator. Patients also receive a booklet entitled, "Cancer Survivorship Next Steps for Patients and Their Families."

After completion of intervention, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of cancer
* Have received surgery, chemotherapy, and/or radiation therapy
* Have completed all surgery, chemotherapy and/or radiation therapy within the last 2-60 months
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-V criteria for insomnia and score >= 10 on the Insomnia Severity Index
* Be able to read and understand English
* Be able to provide written informed consent

Exclusion Criteria:

* Have contraindications to functional testing or yoga participation according to the treating physician
* Have practiced yoga >= 1 day a week within the 3 months prior to enrolling in the study
* Be planning to start yoga on their own during the time they are enrolled in the study
* Have a confirmed diagnosis of sleep apnea or restless leg syndrome
* Be receiving any form of treatment for cancer with the exception of hormonal or biologic therapy
* Have distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mustian, Principal Investigator — University of Rochester NCORP Research Base
Locations (16):
- United States (16):
  - Hawaii MU NCORP, Honolulu, Hawaii
  - Heartland NCORP, Decatur, Illinois
  - Wichita NCORP, Wichita, Kansas
  - Gulf South MU-NCORP, New Orleans, Louisiana
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Metro-Minnesota NCORP, Minneapolis, Minnesota
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - University of Rochester NCORP Research Base, Rochester, New York
  - Southeast Clinical Oncology Research Consortium, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Pacific Cancer Research Consortium Ncorp, Portland, Oregon
  - Greenville Health System NCORP, Greenville, South Carolina
  - Wisconsin NCORP, Marshfield, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Altman BJ, Lin PJ, Mattick LJ, Outland EH, Bautista J, Li CS, Gada U, Morris KM, Knudsen-Clark AM, Mwangi D, DeRollo RE, Kleckner AS, Kleckner IR, Gilmore NJ, Esparaz BT, Curtis A, Conlin A, Monaco G, Hughey JJ, Mustian KM. Blood Clock Correlation Distance (BloodCCD) as a novel marker to detect circadian rhythm disruption in cancer survivors with insomnia. BJC Rep. 2025 Sep 3;3(1):60. doi: 10.1038/s44276-025-00176-9. PMID 40903493

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants were registered but not eligible.
Period: Overall Study
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Started | 251 | 238 | 251
Completed | 185 | 148 | 175
Not Completed | 66 | 90 | 76
Not completed — Other | 19 | 29 | 17
Not completed — Too time consuming | 21 | 26 | 26
Not completed — Withdrawal by Subject | 13 | 18 | 17
Not completed — Medical | 12 | 13 | 9
Not completed — Disliked Study Procedure | 1 | 1 | 4
Not completed — Disliked Intervention | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention) | Total
Number analyzed (Participants) | 251 | 238 | 251 | 740
Age, Continuous [Mean (Full Range); unit: years] | 55 [24 to 85] | 56 [24 to 83] | 57 [28 to 80] | 56 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 216 | 236 | 686
  Male | 17 | 22 | 15 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 5 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 29 | 26 | 28 | 83
  White | 213 | 207 | 214 | 634
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 251 | 238 | 251 | 740
ISI at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index is a validated measure of insomnia. A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia. Population: The difference between the number of participants analyzed and the overall number of baseline participants is due to participant withdrawal.
  units on a scale
    number analyzed (Participants) | 216 | 198 | 205 | 619
    (all) | 15.41 (4.34) | 15.57 (4.35) | 15.39 (4.39) | 15.45 (4.35)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the ISI Comparing YOCAS vs. CBT-I
Description: The Insomnia Severity Index is a validated measure of insomnia. A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia. Means and 95% confidence intervals for YOCAS and CBT-I will be calculated and plotted and examined in comparison with the a priori specified non-inferiority margin of 1.15.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: The overall number of participants analyzed is higher than the number of participants who completed the study because the timeframe for this outcome measure was from baseline up to post-intervention. Some participants withdrew after the post-intervention assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 202 | 163 | 185
units on a scale | -3.61 [-4.19 to -3.03] | -7.22 [-7.95 to -6.49] | -2.19 [-2.84 to -1.55]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); Constructed a 95% confidence interval on the mean change of ISI from baseline between the arms (YOCAS - CBT-I). If the lower bound of the interval is less than 1.5 then we conclude that YOCAS is non-inferior; Test type: Non-Inferiority — Non-inferiority is established if the difference in mean change on the ISI between YOCAS©® and CBT-I is less than 1.15. Using ANCOVA to estimate differences in mean change between YOCAS©® and CBT-I, a correlation of 0.576 (from our prior study), and a sample of 168 subjects per group, we will have sufficient (80%) power to detect non-inferiority using a margin of 1.15 at p = 0.025; p < .0001, Mixed Models Analysis — The p-value shown above is from the Least Squares Mean between YOCAS - CBT-I from the Mixed Model; Mean Difference (Final Values) = 3.52, 95% CI 2-sided [2.66 to 4.37], Standard Error of Mean 0.43 — The comparison is YOCAS - CBT-I

2. Primary Outcome: Mean Change in the ISI Comparing YOCAS vs. Health Education
Description: The Insomnia Severity Index is a validated measure of insomnia. A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 202 | 163 | 185
units on a scale | -3.61 [-4.19 to -3.03] | -7.22 [-7.95 to -6.49] | -2.19 [-2.84 to -1.55]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); The comparison of YOCAS to the health education control is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Superiority — Using ANCOVA to estimate differences in mean change between YOCAS and health education, a correlation of 0.576 (from our prior study), and a sample size of 168 evaluable subjects per group, we will have sufficient power to detect differences on the ISI of at least 1.3, 1.5 and 1.6 (all larger than our 1.15 non-inferiority margin) at 80%, 90%, and 95% power, respectively; p = 0.0009, Mixed Models Analysis — the comparison of YOCAS to the health education control is a traditional null hypothesis of no difference with a two-sided alpha. The p-value shown is from the Least Squares Mean (YOCAS - Health Education) generated from the Mixed Model; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-2.23 to -0.58], Standard Error of Mean 0.42 — The comparison is from the ISI Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

3. Secondary Outcome: Mean Change in Global Sleep Quality Impairment as Measured by the Pittsburgh Sleep Quality Inventory (PSQI) Total Score Comparing YOCAS vs. Health Education
Description: The PSQI measures sleep quality with a total score ranging from 0-21 with higher scores indicating worse sleep quality. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 202 | 163 | 186
units on a scale | -1.59 [-1.99 to -1.18] | -3.82 [-4.30 to -3.33] | -1.11 [-1.55 to -0.68]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.0700, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.98 to 0.04], Standard Error of Mean 0.26 — The comparison is from the ISI Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

4. Secondary Outcome: Mean Change in Global Sleep Quality Impairment as Measured by the Pittsburgh Sleep Quality Inventory (PSQI) Total Score Comparing YOCAS vs. CBT-I.
Description: The PSQI measures sleep quality with a total score ranging from 0-21 with higher scores indicating worse sleep quality. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 202 | 163 | 186
units on a scale | -1.59 [-1.99 to -1.18] | -3.82 [-4.30 to -3.33] | -1.11 [-1.55 to -0.68]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p < .0001, Mixed Models Analysis — The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha. The p-value shown is from the Least Squares Mean (YOCAS - CBT-I) generated from the Mixed Model; Mean Difference (Final Values) = 2.23, 95% CI 2-sided [1.70 to 2.75], Standard Error of Mean 0.27 — The comparison is from the ISI Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

5. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Duration Via Actigraphy Comparing YOCAS vs. Health Education
Description: Actigraphy will measure the number of minutes of actual sleep. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: The overall number of participants analyzed is lower than the number of participants who completed the study. This difference is due to the actigraphy device malfunction or battery issue and participant non-compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 395.99 [383.49 to 408.50] | 380.06 [366.93 to 393.18] | 376.27 [363.06 to 389.48]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.0052, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 19.73, 95% CI 2-sided [5.91 to 33.54], Standard Error of Mean 7.03 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

6. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Duration Via Actigraphy Comparing YOCAS vs. CBT-I
Description: Actigraphy will measure the number of minutes of actual sleep. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 395.99 [383.49 to 408.50] | 380.06 [366.93 to 393.18] | 376.27 [363.06 to 389.48]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.0258, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 15.94, 95% CI 2-sided [1.93 to 29.94], Standard Error of Mean 7.12

7. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Wake After Sleep Onset Via Actigraphy Comparing YOCAS vs. Health Education
Description: Actigraphy will measure total minutes of wake time after sleep onset. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education. The transformation of the log base 10 of the original measurement was used for the analysis.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 1.85 [1.81 to 1.89] | 1.81 [1.76 to 1.85] | 1.86 [1.81 to 1.90]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.053 to 0.048], Standard Error of Mean 0.025 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

8. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Wake After Sleep Onset Via Actigraphy Comparing YOCAS vs. CBT-I
Description: Actigraphy will measure total minutes of wake time after sleep onset. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I. The transformation of log base 10 of the original measurement was used for the analysis.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 1.85 [1.81 to 1.89] | 1.81 [1.76 to 1.85] | 1.86 [1.81 to 1.90]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to the CBT-I control is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.07, Mixed Models Analysis — The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha. The p-value shown is from the Least Squares Mean (YOCAS - Health Education) generated from the Mixed Model; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.004 to 0.098], Standard Error of Mean 0.026 — The comparison is from the Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

9. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Efficiency Via Actigraphy Comparing YOCAS vs. Health Education
Description: Actigraphy will measure the percent of time actually slept compared to intended time sleeping. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of time
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
percent of time | 81.65 [79.57 to 83.73] | 82.42 [80.24 to 84.60] | 79.38 [77.19 to 81.58]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [0.09 to 4.44], Standard Error of Mean 1.11 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

10. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Efficiency Via Actigraphy Comparing YOCAS vs. CBT-I
Description: Actigraphy will measure the percent of time actually slept compared to intended time sleeping. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of time
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
percent of time | 81.65 [79.57 to 83.73] | 82.42 [80.24 to 84.60] | 79.38 [77.19 to 81.58]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.49, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-2.97 to 1.43], Standard Error of Mean 1.12 — The comparison is from the Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

11. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Latency Via Actigraphy Comparing YOCAS vs. Health Education
Description: Actigraphy will measure the minutes it takes for the participant to fall asleep. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and health education. The transformation of log base 10 of the (measurement + 1) was used in the analysis.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 0.76 [0.69 to 0.83] | 0.74 [0.67 to 0.82] | 0.80 [0.73 to 0.87]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.43, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.13 to 0.05], Standard Error of Mean 0.05 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

12. Secondary Outcome: Mean Change in Objective Symptoms of Insomnia- Sleep Latency Via Actigraphy Comparing YOCAS vs. CBT-I
Description: Actigraphy will measure the minutes it takes for the participant to fall asleep. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I. The transformation of the log base 10 of the (measure + 1) was used in the analysis.
Time Frame: Baseline up to post intervention (approximately 4 to 8 weeks)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 150 | 135 | 144
minutes | 0.76 [0.69 to 0.83] | 0.74 [0.67 to 0.82] | 0.80 [0.73 to 0.87]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.70, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.07 to 0.11], Standard Error of Mean 0.05 — The comparison is from the Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

13. Secondary Outcome: Mean Change in the ISI Comparing YOCAS and Health Education (3 Month)
Description: as for outcome 2
Time Frame: Baseline to 3 months
Population: The overall number of participants analyzed in arms I & II is higher than the number of participants who completed the study. This difference is due to some participants withdrew after this outcome measure was collected. The overall number of participants analyzed in arm III is lower than the number of participants who completed the study. This difference is due to participant non-compliance.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 189 | 153 | 173
units on a scale | -5.02 [-5.72 to -4.28] | -7.59 [-8.37 to -6.81] | -3.56 [-4.31 to -2.82]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.0041, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.65 to -0.50], Standard Error of Mean 0.55 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

14. Secondary Outcome: Mean Change in the ISI Comparing YOCAS and CBT-I (3 Month)
Description: The Insomnia Severity Index is a validated measure of insomnia. A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change between YOCAS and CBT-I.
Time Frame: Baseline to 3 months
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 189 | 153 | 173
units on a scale | -5.02 [-5.72 to -4.28] | -7.59 [-8.37 to -6.81] | -3.56 [-4.31 to -2.82]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 2.71, 95% CI 2-sided [1.61 to 3.81], Standard Error of Mean 0.56 — The comparison is from the Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

15. Secondary Outcome: Mean Change in the ISI Comparing YOCAS and Health Education (6 Month)
Description: as for outcome 2
Time Frame: Baseline to 6 months
Population: The overall number of participants analyzed is lower than the number of participants who completed the study. This difference is due to participant non-compliance.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 182 | 144 | 171
units on a scale | -5.29 [-6.00 to -4.57] | -7.93 [-8.71 to -7.15] | -3.91 [-4.75 to -3.07]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm III (Educational Intervention); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p = 0.0108, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.78 to -0.36], Standard Error of Mean 0.62 — The comparison is from the Least Squares Mean difference (YOCAS - Health Education) generated from the Mixed Model

16. Secondary Outcome: Mean Change in the ISI Comparing YOCAS and CBT-I (6 Month)
Description: as for outcome 14
Time Frame: Baseline to 6 months
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
Number analyzed (Participants) | 182 | 144 | 171
units on a scale | -5.29 [-6.0 to -4.57] | -7.93 [-8.71 to -7.15] | -3.91 [-4.75 to -3.07]
Statistical Analysis 1: Comparison: Arm I (Behavioral Intervention-yoga) vs Arm II (Cognitive Intervention-CBT-I); The comparison of YOCAS to CBT-I is a traditional null hypothesis of no difference with a two-sided alpha; Test type: Equivalence — The null hypothesis is that the mean change in the outcome measure between the two arms is zero; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 2.78, 95% CI 2-sided [1.54 to 4.02], Standard Error of Mean 0.63 — The comparison is from the Least Squares Mean difference (YOCAS - CBT-I) generated from the Mixed Model

ADVERSE EVENTS:
Time Frame: 1 year and 9 months
Arm/Group | Arm I (Behavioral Intervention-yoga) | Arm II (Cognitive Intervention-CBT-I) | Arm III (Educational Intervention)
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/238 | 0/251
Serious Adverse Events (participants affected / at risk) | 3/251 | 1/238 | 1/251
Other Adverse Events (participants affected / at risk) | 0/251 | 0/238 | 0/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Behavioral Intervention-yoga) (N=251) | Arm II (Cognitive Intervention-CBT-I) (N=238) | Arm III (Educational Intervention) (N=251)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Confusion/brain met (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage/brain met (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intraparenchymal hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT02613364/Prot_SAP_000.pdf